CLINICAL TRIAL: NCT06091670
Title: Genital Hygiene Behaviors and Predicting Factors in Women Living in A Country: The Sample of Turkey
Brief Title: Genital Hygiene Behaviors and Predicting Factors
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esra Çalışkan, Phd Student, Istanbul University - Cerrahpasa
Other Study IDs: ECaliskan1
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Urinary Tract Infections
Keywords: genital hygiene; female genital; hygiene behaviour; women's health
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention. The research is cross-sectional-descriptive type.

SUMMARY:
The aim of this study was to determine the genital hygiene practices of women in different regions of Turkey and the factors influencing these practices. It is a descriptive, cross-sectional study. The study was conducted according to the STROBE checklist.

DETAILED DESCRIPTION:
The aim of this study was to determine the genital hygiene practices of women in different regions of Turkey and the factors influencing these practices. It is a descriptive, cross-sectional study.

Data Collection Tools Data for the study was collected through the "Data Collection Form" and "Genital Hygiene Behaviors Inventory", created by the researchers by reviewing the literature (Karahan, 2017; Cankaya, 2013; Elzayat et al. 2017; Adam and Saadia, 2016; Akgul, 2019).

Data collection form: A survey consisting of 13 questions about the age of the women, the amount of water consumed daily, the number of urinations, the genital infection status, and sexuality.

Genital Hygiene Behaviors Inventory - GHBI: A scale, developed by Karahan (2017), and for which written permission for use was obtained, consisting of 23 items in total and 3 sub-dimensions: "genital hygiene behaviors", "menstrual habits" and "abnormal findings". Items 1-12 evaluate genital hygiene, items 13-20 evaluate menstrual hygiene, and items 21-23 evaluate the awareness of abnormal findings. Items 7, 14, 19, 20 and 23 of the scale are the reversed items and are reverse coded during the evaluation. A minimum total of 23 and a maximum total of 115 points can be obtained from the 5-point Likert-type scale, where "1" point means "I totally disagree" and "5" points means "I completely agree". Higher scale scores correspond to better genital hygiene behaviors. The study evaluating the development of the scale and its validity and reliability determined the Cronbach's Alpha coefficient as 0.80 (Karahan, 2017); our study's Cronbach's Alpha coefficient was 0.78.

Data Collection The prepared data collection form and the scale were transferred to the computer environment and delivered online to the women through the snowball sampling method. It took approximately 10 minutes for each participant to complete the data collection forms Data Analysis The data collected in the study was analyzed using the Statistical Package for the Social Sciences, version 25.0 (SPSS, v25.0) statistical analysis package program (IBM Company, Turkey). First the descriptive data of the study was analyzed. Mean, median, standard deviation, minimum and maximum values were calculated in the analysis of continuous data, and numbers and percentages were calculated in the analysis of categorical data. Next, non-parametric and parametric tests were used according to normality distributions. Pearson Chi-square test, Kruskal Wallis Test and Mann Whitney-U tests were used to analyze the data. A simple linear regression analysis model was used to determine the factors affecting genital hygiene behaviors. Statistical significance level was accepted as p<.05 at 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study,
* To speak and understand Turkish,
* women

Exclusion Criteria:

* not being able to read and understand Turkish
* dont want to participate the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of all women throughout Turkey, while the sample consisted of women who met the inclusion criteria of the study.
  The criteria for inclusion in the study are: (i) being able to read and understand Turkish, (ii) meeting the conditions for voluntary participation in the study. The sample consisted of 881 women reached online by the snowball sampling method
Sampling Method: Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Genital Hygiene Behavior Inventory (GHBI) | 1 times
  Likert type inventory consisting of 27 questions evaluating genital hygiene behaviors.Inventory was applied to all pregnant women participating in the study at the beginning and at the end of the study.
Data collection form: | 1 times
  This survey was created by the researchers according to the literature.6-9 The survey consisted of 13 questions about the sociodemographic features and the behaviors related genital tract infections.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Çalışkan, Msc, Study Director — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No
Research results will be shared

REFERENCES:
- [Background] Emiru T, Beyene G, Tsegaye W, Melaku S. Associated risk factors of urinary tract infection among pregnant women at Felege Hiwot Referral Hospital, Bahir Dar, North West Ethiopia. BMC Res Notes. 2013 Jul 25;6:292. doi: 10.1186/1756-0500-6-292. PMID 23885968
- [Background] Minardi D, d'Anzeo G, Cantoro D, Conti A, Muzzonigro G. Urinary tract infections in women: etiology and treatment options. Int J Gen Med. 2011;4:333-43. doi: 10.2147/IJGM.S11767. Epub 2011 Apr 19. PMID 21674026
- [Background] Abdel-Aziz Elzayat M, Barnett-Vanes A, Dabour MF, Cheng F. Prevalence of undiagnosed asymptomatic bacteriuria and associated risk factors during pregnancy: a cross-sectional study at two tertiary centres in Cairo, Egypt. BMJ Open. 2017 Mar 21;7(3):e013198. doi: 10.1136/bmjopen-2016-013198. PMID 28325856
- [Background] Haider G, Zehra N, Munir AA, Haider A. Risk factors of urinary tract infection in pregnancy. J Pak Med Assoc. 2010 Mar;60(3):213-6. PMID 20225781
- [Background] Stapleton A, Stamm WE. Prevention of urinary tract infection. Infect Dis Clin North Am. 1997 Sep;11(3):719-33. doi: 10.1016/s0891-5520(05)70382-2. PMID 9378932